CLINICAL TRIAL: NCT00026260
Title: A Phase II Evaluation of SU5416 (NSC 696819) in Persistent or Recurrent Squamous Cell Carcinoma of the Cervix
Brief Title: SU5416 in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069013; GOG-0227B
Record Dates: First submitted 2001-11-09; First posted 2003-10-21 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2007-06

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Semaxinib

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
RATIONALE: Biological therapy with drugs such as SU5416 may stop the growth of cervical cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of SU5416 in treating patients who have persistent or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor cytostatic activity of SU5416, in terms of 6-month progression-free survival and time to progression, in patients with persistent or recurrent cervical squamous cell carcinoma.
* Determine the nature and degree of toxicity of this drug in these patients.
* Correlate surrogate endpoint molecular and imaging markers with clinical outcome in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive SU5416 IV over 1 hour on days 1 and 4. Treatment repeats weekly in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 19-51 patients will be accrued for this study within 8-23 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cervical squamous cell carcinoma

  * Persistent or recurrent disease with documented progression
  * No nonsquamous cell cervical malignancies, including adenosquamous carcinoma
* At least 1 measurable lesion

  * At least 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI OR
  * At least 10 mm by spiral CT scan
* Failed prior local therapeutic measures
* Ineligible for higher priority GOG protocol (e.g., any active GOG phase III protocol for the same patient population)
* Tumor must be accessible for biopsy using direct- or guided-needle technique

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least lower limit of normal
* Absolute neutrophil count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No uncompensated coronary artery disease on electrocardiogram or physical examination
* No myocardial infarction within the past 6 months
* No severe/unstable angina within the past 6 months
* No severe peripheral vascular disease
* No deep vein or arterial thrombosis within the past 3 months

Pulmonary:

* No pulmonary embolism within the past 3 months

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Must have central venous access
* No uncontrolled diabetes mellitus
* No prior allergic reaction to paclitaxel
* No active infection requiring antibiotics
* No peripheral neuropathy greater than grade 1
* No contraindications to low-dose (1 mg/day) warfarin or low-molecular weight heparin prophylaxis
* No claustrophobia that would preclude MRI studies
* No ferromagnetic implants or pacers
* No other invasive malignancy within the past 5 years except non-melanoma skin cancer
* No other concurrent circumstances that would preclude study completion

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Biologic therapy:

* No prior antiangiogenesis agents, including SU5416
* At least 3 weeks since prior biologic or immunologic agents directed at malignancy

Chemotherapy:

* No more than 1 prior chemotherapy regimen, including single or combination cytotoxic drug therapy (radiosensitizers do not count as prior regimen)
* At least 3 weeks since prior chemotherapy directed at malignancy and recovered

Endocrine therapy:

* At least 1 week since prior hormonal therapy directed at malignancy
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* At least 3 weeks since prior radiotherapy directed at malignancy and recovered

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior surgery for malignancy and recovered

Other:

* No prior cancer therapy that would preclude study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Burger, MD, Study Chair — Chao Family Comprehensive Cancer Center